CLINICAL TRIAL: NCT01501240
Title: Gadoxetic Acid-enhanced MR Evaluation of Hepatocellular Carcinoma and Dysplastic Nodules in the Cirrhotic Liver: Prospective Pathologic Correlation With Explanted Liver
Brief Title: Gadoxetic Acid-enhanced MR Evaluation of Hepatocellular Carcinoma and Dysplastic Nodules in the Cirrhotic Liver
Acronym: PriMPa
Status: Withdrawn | Type: Observational
Sponsor: Jae Ho Byun (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, Jae Ho Byun, Associate Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMC-2011-0797
Record Dates: First submitted 2011-12-26; First posted 2011-12-29 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Liver Cirrhosis; Carcinoma, Hepatocellular
Keywords: Magnetic resonance image; gadoxetic acid; hepatocellular carcinoma; liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- liver cirrhosis, liver transplantation: Patients with known liver cirrhosis and planned to undergo liver transplantation within 1 month will be eligible population in the study

SUMMARY:
A prospective intra-individual study to investigate the diagnostic performance of gadoxetic acid-enhanced MR for the patients with liver cirrhosis using thin-section whole-explant as standard of reference

DETAILED DESCRIPTION:
Liver cirrhosis is a progressive, diffuse disease of the liver characterized by hepatocyte necrosis, fibrosis, distortion of the normal hepatic architecture and a spectrum of nodular lesions that includes regenerative nodules (RN), dysplastic nodules (DN) and hepatocellular carcinomas (HCC). Since HCC is the leading cause of death among the patients with liver cirrhosis, Early and accurate diagnosis of HCC and its precursors by using optimal imaging technique is critical for its treatment and management.

Recently state-of-the-art magnetic resonance (MR) imaging with gadoxetic acid, which works both an extracellular and hepatocyte-specific contrast agent, has been increasing used to evaluate the patients with liver cirrhosis. Several studies correlated gadoxetic acid-enhanced MR of HCC and hepatocellular nodules with the pathology from biopsy or surgical resection specimens. However, all of those studies are limited by its lack of complete correlation between pathologic and imaging findings and the resulting bias being toward the positive studies. Ideally, the use of whole explant pathologic correlation would be helpful for exact characterization of HCC and its precursors on gadoxetic acid-enhanced MR.

The question of our study is how accurate gadoxetic acid-enhanced MR is in the evaluation of the patients with cirrhotic liver to detect HCC and dysplastic nodules and, by using thin-section whole-explant correlation following liver transplantation as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known liver cirrhosis based on either histology, or a combination of physical examination, laboratory tests, and imaging data
* Patients with known liver cirrhosis based on either histology, or a combination of physical examination, laboratory tests, and imaging data

Exclusion Criteria:

* Patients under 20 years of age
* Patients who have more than 10 nodules detected on hepatobiliary phase of gadoxetic acid-enhanced MR
* Patients who underwent transarterial chemotherapy or radiofrequency ablation
* Women who are pregnant, lactating or who are of childbearing potential
* Patients with any physical or mental status than interferes with the signing of informed consent
* Patients with a contraindication for MR
* Patients with impaired renal function (e.g. acute renal failure or eGFR < 30 ml/min/1.73m2) or patients on dialysis

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known liver cirrhosis and planned to undergo liver transplantation within 1 month
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Diagnostic sensitivity of gadoxetic acid-enhanced MR imaging to detect HCC in the cirrhotic liver, using thin-section whole-explant as the standard of reference | Within the first week after liver explantation

SECONDARY OUTCOMES:
Specificity of gadoxetic acid-enhanced MR imaging to detect HCC in the cirrhotic liver, using thin-section whole-explant as standard of reference | Within the first week after liver explantation
Sensitivity and specificity of gadoxetic acid-enhanced MR imaging to detect dysplastic nodules | Within one week after liver transplantation
  To assess the diagnostic sensitivity and specificity of gadoxetic acid-enhanced MR imaging to detect dysplastic nodules in the cirrhotic liver, using thin-section whole-explant as standard of reference
To characterize borderline hepatocelluar nodules | Within one week after liver transplantation
  To characterize borderline hepatocelluar nodules (i.e.,1-3cm sized nodules without arterial hypervascularity) in the cirrhotic liver detected on hepatobiliary phase of gadoxetic acid-enhanced MR

CONTACTS AND LOCATIONS:
Overall Officials: Jae Ho Byun, MD, PhD, Principal Investigator — University of Ulsan College of Medicine, Asan Medical Center
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - Division of Abdomen, Department of Radiology & Research Institute of Radiology, University of Ulsan College of Medicine, Asan Medical Center, Seoul

REFERENCES:
- [Background] Kudo M. Will Gd-EOB-MRI change the diagnostic algorithm in hepatocellular carcinoma? Oncology. 2010 Jul;78 Suppl 1:87-93. doi: 10.1159/000315235. Epub 2010 Jul 8. PMID 20616589
- [Background] Zech CJ, Reiser MF, Herrmann KA. Imaging of hepatocellular carcinoma by computed tomography and magnetic resonance imaging: state of the art. Dig Dis. 2009;27(2):114-24. doi: 10.1159/000218343. Epub 2009 Jun 22. PMID 19546549
- [Background] Tanimoto A, Lee JM, Murakami T, Huppertz A, Kudo M, Grazioli L. Consensus report of the 2nd International Forum for Liver MRI. Eur Radiol. 2009 Oct;19 Suppl 5:S975-89. doi: 10.1007/s00330-009-1624-y. PMID 19851766